



## STROKE PARTICIPANT CONSENT FORM

Study title: Identifying vertical perception loss in people with acute stroke. A feasibility study.

Researchers: Amelia Shaw, Dr. Katherine Cook, Dr. Louise Johnson and Dr. James Faulkner

IRAS ID: 333405

Participant Identification Number for this trial:

You are consenting to participate in a research study through the completion of three assessments:

- Assessments one and two involve a therapist watching you do some activities and recording the results.
- For assessment three you will sit and look inside a bucket and tell the assessor when the line on the bottom of the bucket is vertical.

This research wants to establish if it is possible to do these assessments soon after having a stroke.

## Please <u>initial</u> the boxes if you agree with the statements:

| I have read and understood participant information sheet version 2 dated 24/1/24 and have had the opportunity to ask questions about the study. |
|---|
| I agree to take part in this research project and agree for my data to be used for the purpose of this study. |
| I understand my participation is voluntary and I can withdraw at any point until I am discharged from the stroke unit and this will not impact my ongoing care. Any data from assessments completed prior to my withdrawal will be used in the results but will be anonymous. |
| I agree that anonymised data can be accessed by researchers not involved in this study for use in secondary data analysis. |
| I understand that my medical record may be accessed by appropriately qualified people from Hampshire<br>Hospitals NHS Foundation Trust in relation to this research |

Version 2 24/1/24 IRAS ID: 333405





| I agree to have the three assessments repeated at the end of my admission, but understand that this will not apply to all participants. |
|---|
| I agree to participate in a survey when I have completed the assessments or at four weeks after agreeing to participate in the study, whichever is the soonest. |
| I agree to participate in this study |
| Name of participant (print name) |

When completed: 1 (original) to be kept in care record, 1 for consultee; 1 for researcher site file

Signature of researcher ......Date.......Date.....

Signature of participant......Date: ......Date:

Name of researcher (print name).....

Version 2 24/1/24

IRAS ID: 333405